CLINICAL TRIAL: NCT01093378
Title: Impact of the Diet Fertility : A Case-control Multicentric Study
Brief Title: Diet and Its Relationship With Couple Infertility
Acronym: ALIFERT
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University Paris 7 - Denis Diderot (Other)
Responsible Party: Sponsor
Other Study IDs: P071224
Record Dates: First submitted 2010-02-26; First posted 2010-03-25 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Infertility
Keywords: Infertility; Obesity; Dietary intake; Fertility; nutrition; diet; weight
MeSH Terms: conditions — Infertility; Obesity; Body Weight

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Impact of genetic polymorphism on clinical and biological phenotypes linked to food behaviour in infertility context
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fertile group: fertile group
- Infertility group: Fertility troubles

SUMMARY:
This case-control multicentric study involving fertile and infertile couples aims at evaluating the impact on conception rate of nutritional parameters (biologic, clinic, anthropometric, and food questionnaire).

DETAILED DESCRIPTION:
Infertility affects about 15% of couples. Many factors relating to lifestyle and environment are likely to influence fertility. As an adapted nutrition could prevent 30% of cancers, diet could be essential, but largely neglected, in the prevention of infertility.

Some studies tried to explore the impact of diet on male or female fertility, but very few focused on both. The aim of our study is to assess the role of nutrition in both fertile and infertile couples, taking into account most of factors relating to lifestyle. Clinical, anthropometric (BMI, fat mass), biological markers (non specific - glycaemia, lipids, inflammation, electrolytes - and specific - vitamins E, A, C, D, B, including folates and MTHFR polymorphism) and semen analysis, will be combined with validated questionnaires (nutrition, drugs, alcohol, tobacco, physical activity, sleep and stress).

The statistical analysis of correlations between nutritional and clinical data will provide information concerning the impact of nutrition on fertility.

ELIGIBILITY:
Inclusion Criteria:

Common to both infertile and fertile couples:

* Couples where both members are over eighteen and at childbearing age (≤38 for women and ≤ 45 for men)
* Couples where both members agreed to take part in the study
* Couples where both members completed a medical check-up and gave an informed consent. Infertile couples could be included following a medical consultation for infertility
* Couples with none of its member facing any comprehension difficulty in oral or written French language
* Couples where both members are affiliated to the French NHS [national health service] (beneficiary or legal claimant)

Specific to fertile couples:

- fertile couples who naturally and spontaneously conceived a or many children with a time to conceive shorter than 12 months.

Specific to infertile couples:

* Infertile couples (primary, infertility, inability to conceive a child after 12 months of unprotected sexual intercourse)
* Couples where the male partner has sperm parameters compatible with a natural conception
* Couples where the female partner does not present anovulation, ovarian insufficiency and or any uterus-tubal pathology

Exclusion Criteria:

Common to both infertile and fertile couples:

* couples where one of the members is under eighteen or not a childbearing age (>38 for women an >45 for men)
* couples where at least one member refused to give written agreement for the study
* couples where at least one member shows any known cardiovascular risk (diabetes, hypercholesterolemia, HBR)
* couples where at least one member shows any known cardiovascular pathology, digestive pathology, no good absorptive pathology or a cancer
* couples where at least one member faces some difficulty in understanding French language
* couples where at least one member is not affiliated with the French NHS (beneficiary or legal claimant)

Specific to fertile couples:

•Couples where the woman had a miscarriage or medical termination of pregnancy with current partner

Specific to infertile couples:

* Couples in which it is not the first pregnancy
* Couples with the male member showing either:

  * severe oligozoospermia (<5 millions/ml) or a confirmed azoospermia (absence of spermatozoid in the ejaculate)
  * a moderate non idiopathic oligozoospermia (5-20 millions/ml), related to one more of the following factors:

    1. toxic (chemotherapy, radiotherapy, drugs with a demonstrated effect on spermatogenesis)
    2. infectious
    3. anatomic: vasectomy, congenital anomaly (agenesis of vas deferens), long post-traumatic ischemia
    4. endocrine: hypogonadotropic, hypogonadism
    5. cytogenetic: klinefelter syndrome, translocation
* couples whose male partner shows an abnormality of the male genital tractus : VARICOCEME undescended,testis, testicular volume < 12ml
* couples whose female partner presents an anovulation, ovarian insufficiency or a proven uterus-tubal pathology

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Defined population after a screening in out-hospitalized patients in selected investigation sites
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2009-10; Primary Completion 2013-10 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the nutritional status of fertile and infertile couples (food questionnaire - biologic, anthropometric and clinical balance). | 24 hours

SECONDARY OUTCOMES:
Impact of genetic polymorphism on clinical and biological phenotypes linked to food behaviour in infertility context (MTHFR polymorphism for folates metabolism) | 12 months
Impact of lifestyle (alcohol and tabacco consumption, physical activity, anxiety and sleep) on diet and fertility | 24 hours
Impact of nutritional status on fertility and ART parameters | 24 hours
Fertility : time to pregnancy (TTP) | in the 6 months
Male infertility : quantitative or qualitative semen abnormalities | in the 6 months
Pregnancy and obstetrical pathologies, prematurity, twin birth, weight of the new-born in infertile couples | in the 6 months
ART parameters, if appropriate | in the 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Levy, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Laboratoire d'Histologie- Embryologie - Cytogénétique - CECOS, Bondy, France

REFERENCES:
- [Derived] Caetano G, Rouen A, Dupont C, Levy R, Leger D, Sermondade N; ALIFERT Collaborative Group. Sleep and idiopathic infertility: a case-control study of 360 participants. Reprod Biomed Online. 2025 Nov;51(5):105040. doi: 10.1016/j.rbmo.2025.105040. Epub 2025 May 7. PMID 40865394
- [Derived] Bachelot G, Levy R, Bachelot A, Faure C, Czernichow S, Dupont C, Lamaziere A; Alifert Collaborative Group. Proof of concept and development of a couple-based machine learning model to stratify infertile patients with idiopathic infertility. Sci Rep. 2021 Dec 14;11(1):24003. doi: 10.1038/s41598-021-03165-3. PMID 34907216
- [Derived] Talla P, Faure C, Rigourd V, Czernichow S, Sermondade N, Levy R, Dupont C; ALIFERT collaborative group. Is There an Association of Being Breastfed as an Infant and Fertility Status as an Adult? Breastfeed Med. 2021 May;16(5):414-418. doi: 10.1089/bfm.2020.0130. Epub 2021 Mar 30. PMID 33781087
- [Derived] Dupont C, Hulot A, Jaffrezic F, Faure C, Czernichow S, di Clemente N, Racine C, Chavatte-Palmer P, Levy R; Alifert group. Female ponderal index at birth and idiopathic infertility. J Dev Orig Health Dis. 2020 Apr;11(2):154-158. doi: 10.1017/S2040174419000394. Epub 2019 Jul 16. PMID 31309911
- [Derived] Dupont C, Faure C, Daoud F, Gautier B, Czernichow S, Levy R; ALIFERT collaborative group. Metabolic syndrome and smoking are independent risk factors of male idiopathic infertility. Basic Clin Androl. 2019 Jul 1;29:9. doi: 10.1186/s12610-019-0090-x. eCollection 2019. PMID 31304019
- [Derived] Faure C, Dupont C, Chavatte-Palmer P, Gautier B, Levy R; ALIFERT Collaborative Group. Are semen parameters related to birth weight? Fertil Steril. 2015 Jan;103(1):6-10. doi: 10.1016/j.fertnstert.2014.11.027. PMID 25552408
- [Derived] Faure C, Leveille P, Dupont C, Julia C, Chavatte-Palmer P; Alifert Group; Sutton A, Levy R. Are superoxide dismutase 2 and nitric oxide synthase polymorphisms associated with idiopathic infertility? Antioxid Redox Signal. 2014 Aug 1;21(4):565-9. doi: 10.1089/ars.2014.5831. Epub 2014 Feb 25. PMID 24444339